CLINICAL TRIAL: NCT00651144
Title: SCH 058235: Assessment of a Multiple-Dose Drug Interaction Between Ezetimibe and Rosuvastatin in Healthy Hypercholesterolemic Subjects
Brief Title: Assessment of Potential Interaction Between Ezetimibe and Rosuvastatin in Healthy Subjects With High Cholesterol (P03317)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P03317
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Atherosclerosis
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ezetimibe + Rosuvastatin (Experimental)
  Interventions: Drug: Ezetimibe + Rosuvastatin
- Ezetimibe (Active Comparator)
  Interventions: Drug: Ezetimibe
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezetimibe + Rosuvastatin — oral tablets; rosuvastatin 10 mg + ezetimibe 10 mg, once daily for 14 days
  Other Names: Zetia; SCH 58235; Crestor
  Arms: Ezetimibe + Rosuvastatin
Drug: Rosuvastatin — oral tablets; rosuvastatin 10 mg + ezetimibe placebo once daily for 14 days
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Placebo — oral tablets; two ezetimibe placebo once daily for 14 days
  Arms: Placebo
Drug: Ezetimibe — oral tablets; ezetimibe 10 mg + ezetimibe placebo once daily for 14 days
  Other Names: Zetia; SCH 58235
  Arms: Ezetimibe

SUMMARY:
The purpose of this study is to obtain data of the coadministration of ezetimibe and rosuvastatin to support the concomitant use of these two drugs in patients requiring additional cholesterol-lowering management. Treatment is administered for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 55 years inclusive, having a Body Mass Index (BMI) between 19-31 inclusive. BMI=weight (kg)/height (m^2).
* Subjects must have untreated hypercholesterolemia with a directly measured fasting LDL-C >=130 mg/dL (3.37 mmol/L) at Screening and on Day -1. Subjects must be free of any clinically significant disease that requires a physician's care and/or would interfere with the study evaluations.
* Subjects must have a normal or clinically acceptable physical exam and ECG (12-lead recorded at 25 mm/s and reporting heart rate and PR, QRS, QT, and QTc intervals).
* Subjects' clinical laboratory tests (CBC, blood chemistries, and urinalysis) must be within normal limits or clinically acceptable to the investigator/ sponsor.
* Screen for drugs with high potential for abuse must be negative.
* Subjects must be willing to give written informed consent and able to adhere to dose and visit schedules.
* Subjects must be willing to comply with the NCEP Step 1 diet for at least one week as outpatients, and during the inpatient treatment period.
* Female subjects must be of nonchildbearing potential (ie, surgically sterilized or postmenopausal for at least one year), or, if they are of childbearing potential they must be using a medically accepted method of birth control prior to Screening and agree to continue its use during the study or be surgically sterilized (eg, hysterectomy or tubal ligation). Females of childbearing potential should be counseled in the appropriate use of birth control while in this study. Females who are not currently sexually active must agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the study.
* Female subjects must have a negative serum pregnancy test (beta-hCG) at Screening.

Exclusion Criteria:

* Female subjects who are pregnant, intend to become pregnant, or are nursing.
* Subjects who previously received or were treated with ezetimibe (SCH 58235) or rosuvastatin.
* Subjects who previously received or were treated with lipid lowering drugs (including OTC fish oil and phytosterols) within 6 weeks of Visit 1.
* Any subject who does not comply with the requirement that he/she should not have used any prescription or over-the-counter drugs (except for aspirin or acetaminophen [paracetamol]) within two weeks prior to study drug administration nor alcohol within 48 hours prior to study drug administration.
* Subjects who have used any investigational drugs or donated blood within 30 days of study entry.
* Subjects with pre-existing gallbladder disease or a history of liver function test abnormalities.
* Subjects who smoke more than ten cigarettes or equivalent tobacco use per day.
* Subjects who have a clinically significant allergy or intolerance to foods or drugs, especially to any component of ezetimibe (ZETIA™/EZETROL™) or rosuvastatin (CRESTOR™).
* Subjects who are positive for HIV antibodies, hepatitis B surface antigen or hepatitis C antibody.
* Subjects with a history of mental instability or who have been or are being treated for mood disorders.
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Subjects who are participating in any other clinical study.
* Subjects who are part of the staff personnel directly involved with this study.
* Subjects who are a family member of the investigational study staff.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-03; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in total cholesterol, LDL-C, HDL-C, and triglycerides. | Day 15
Safety: adverse events, laboratory test results, physical examination, vital signs. | Throughout study

SECONDARY OUTCOMES:
Evaluate potential for PK interaction between ezetimibe and rosuvastatin as indicated by Cmax and AUC. | Day 14

REFERENCES:
- [Result] Kosoglou T, Statkevich P, Yang B, Suresh R, Zhu Y, Boutros T, Maxwell SE, Tiessen R, Cutler DL. Pharmacodynamic interaction between ezetimibe and rosuvastatin. Curr Med Res Opin. 2004 Aug;20(8):1185-95. doi: 10.1185/030079904125004213. PMID 15324521